CLINICAL TRIAL: NCT04999436
Title: APOL1 Genetic Testing Program for Living Donors, Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Principal Investigator, Elisa Gordon, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: R01 DK128207 part 2; R01DK128207 (NIH)
Record Dates: First submitted 2021-05-11; First posted 2021-08-10 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Diseases; Genetic Predisposition
Keywords: Implementation science; Ethics; African continental ancestry group; Culturally competent care; Shared decision making; Genetic couseling; Informed consent; Nephrology; Educational intervention; Surveys and questionnaires; Apolipoprotein L1
MeSH Terms: conditions — Renal Insufficiency, Chronic; Genetic Predisposition to Disease

STUDY DESIGN:
Intervention Model Description: We will collect observational data to assess the impact of the training program on clinical practice. We will collect pre-test data before the intervention, and post-test data after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Counseling Training Program (Experimental): The APOL1 counseling training program is designed for transplant nephrologists who evaluate live kidney donor candidates of African ancestry who are at risk for having APOL1 risk variants and kidney failure post-donation. The training program aims to increase transplant nephrologists' practical knowledge, self-efficacy, and skills in counseling live donor candidates about APOL1 in a culturally competent manner. The program will include training in: current APOL1 data; the value of APOL1 testing and meaning of positive test results for living donor clinical evaluation; risks of having two APOL1 gene variants on the donor's kidney health; how to engage in shared decision making about donation; how to address cultural concerns about genetic testing; and how to protect donor candidates' privacy and confidentiality with APOL1 test results. The APOL1 counseling training program will be delivered by a genetic counselor through webinars and other interactive modalities and last 2-4 hours.
  Interventions: Behavioral: APOL1 Counseling Training Program

INTERVENTIONS:
Behavioral: APOL1 Counseling Training Program — The APOL1 counseling training program is designed for transplant nephrologists who evaluate live kidney donor candidates of African ancestry who are at risk for having APOL1 risk variants and kidney failure post-donation. The training program aims to increase transplant nephrologists' practical knowledge, self-efficacy, and skills in counseling live donor candidates about APOL1 in a culturally competent manner. The program will include training in: current APOL1 data; the value of APOL1 testing and meaning of positive test results for living donor clinical evaluation; risks of having two APOL1 gene variants on the donor's kidney health; how to engage in shared decision making about donation; how to address cultural concerns about genetic testing; and how to protect donor candidates' privacy and confidentiality with APOL1 test results. The APOL1 counseling training program will be delivered by a genetic counselor through webinars and other interactive modalities and last 2-4 hours.

SUMMARY:
Living donor (LD) kidney transplantation is the optimal treatment for patients with end-stage kidney disease (ESKD). However, LDs take on a higher risk of future ESKD themselves. African American (AA) LDs have an even greater, 3.3-fold, risk of ESKD than white LDs post-donation. Because evidence suggests that Apolipoprotein L1 (APOL1) risk variants contribute to this greater risk, transplant nephrologists are increasingly using APOL1 testing to evaluate LD candidates of African ancestry. However, nephrologists do not consistently perform genetic counseling with LD candidates about APOL1 due to a lack of knowledge and skill in counseling about APOL1. Without proper counseling, APOL1 testing will magnify LD candidates' decisional conflict about donating, jeopardizing their informed consent. Given their elevated risk of ESRD post-donation, and AAs' widely-held cultural concerns about genetic testing, it is ethically critical to protect AA LD candidates' safety through APOL1 testing in a culturally competent manner to improve informed decisions about donating.

No transplant programs have integrated APOL1 testing into LD evaluation in a culturally competent manner. Clinical "chatbots," mobile apps that use artificial intelligence to provide genetic information to patients and relieve constraints on clinicians' time, can improve informed treatment decisions and reduce decisional conflict. The chatbot "Gia," created by a medical genetics company, can be adapted to any condition. However, no chatbot on APOL1is currently available. No counseling training programs are available for nephrologists to counsel AA LDs about APOL1 and donation in a culturally competent manner. Given the shortage of genetic counselors, increasing nephrologists' genetic literacy is critical to integrating genetic testing into practice.

The objective of this study is to culturally adapt and evaluate the effectiveness of an APOL1testing program for AA LDs at two transplant centers serving large AA LD populations (Chicago, IL, and Washington, DC). The APOL1 testing program will evaluate the effect of the culturally competent testing, chatbot, and counseling on AA LD candidates' decisional conflict about donating, preparedness for decision-making, willingness to donate, and satisfaction with informed consent. The specific aims are to:

1. Adapt Gia and transplant counseling to APOL1 for use in routine clinical practice
2. Evaluate the effectiveness of this intervention on decisional conflict, preparedness, and willingness to donate in a pre-post design
3. Evaluate the implementation of this intervention into clinical practice by using the RE-AIM framework to longitudinally evaluate nephrologist counseling practices and LDs' satisfaction with informed consent.

The impact of this study will be the creation of a model for APOL1 testing of AA LDs, which can then be implemented nationally via implementation science approaches. APOL1 will serve as a model for integrating culturally competent genetic testing into transplant and other practices to improve patient informed consent.

DETAILED DESCRIPTION:
Clinical practice guidelines advise "…considering APOL1 genotyping in live kidney donor candidates with sub-Saharan African ancestors" and using shared decision making until the NIH APOLLO study of APOL1 outcomes in living donors provides population-level data. Transplant physicians are increasingly adopting APOL1 testing. However, physicians do not consistently inform live donor candidates about APOL1, perform genetic counseling, or practice shared decision making with live donor candidates. Our prior research has shown that this variation results from lack of knowledge and skill in counseling about APOL1, and fear that APOL1 testing will deter live donor candidates from donating. It is unknown if they address African American live donor candidates' cultural concerns about genetic testing while counseling.

Effective counseling about APOL1 test results is critical especially because genetic information can magnify live kidney donor candidates' decisional conflict about donating. The consequences of such decisional conflict may be reduced donation rates, which could exacerbate disparities in African Americans patients' access to living donor kidney transplants and health outcomes. Therefore, effective culturally competent counseling is ethically essential to reduce live donor candidates' decisional conflict and enable informed decisions about donation.

This project will entail adapting established genetic counseling discussions for transplant nephrologists to counsel donor candidates about APOL1 test results and engage in shared decision making to improve live donor candidates' informed consent for living donation. The APOL1 counseling training program will address nephrologists' practical knowledge and counseling skill deficits about APOL1 as identified in our prior work. The specific duration and format of the counseling training program will be finalized through a final nephrologist needs assessment early in Year 1. Our preliminary needs assessment revealed a preference for a 2-4 hour educational program delivered by a genetics counselor through a live webinar format. The investigators plan to enroll all transplant nephrologists who evaluate live kidney donor candidates (n=6) across both sites for participation in the counseling training program.

The effectiveness of the nephrologist counseling training program will be assessed primarily by assessing increases in nephrologists' skill in delivering counseling for APOL1 by comparing the number and quality of prescribed counseling behaviors observed between nephrologists counseling live donor candidates in the control group (year 1) versus intervention group (years 2-5). Secondarily, we will evaluate the counseling training program via paired tests of pre-post scores of validated surveys assessing practical knowledge and skills in counseling. Additionally, we will qualitatively analyze nephrologists' perceptions of their APOL1 counseling over time.

Training materials will be updated after two years of implementing the APOL1 intervention based on lessons learned, and will be available for future dissemination. The findings generated from this research have the potential to meaningfully protect donor candidate safety by providing culturally competent counseling and shared decision making to improve candidates' informed consent. As such, we believe this proposal is both timely and responsive to the NIDDK Program Announcement (PA-18-330) "Investigator-Initiated Clinical Trials Targeting Diseases within the Mission of NIDDK."

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years and older)
* English-speaking
* Transplant nephrologists evaluating live kidney donor candidates practicing at the study sites
* Not vision impaired
* Not cognitively impaired

Exclusion Criteria:

* Not a nephrologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Number and quality of prescribed Pre-Test counseling practices | Post-intervention, up to 5 years
  We will use an observer checklist to directly observe participating nephrologists' counseling discussions with live donor kidney transplant candidates' about APOL1 testing, and living donation (before APOL1 testing is done). The checklist will assess the presence/absence of prescribed counseling practices (fidelity) and a rating of each practice's quality (excellent, very good, good, fair, poor).
  The fidelity minimum and maximum values are: 0-12 Higher fidelity scores mean that the pre-test counseling discussion exhibited greater fidelity (adherence) to the training program.
  The quality minimum and maximum values are: 1-5 Higher quality scores mean a better quality counseling discussion.
Number and quality of prescribed Post-Test counseling practices | Post-intervention, up to 5 years
  We will use an observer checklist to directly observe participating nephrologists' counseling discussions with live donor candidates' about APOL1 test results and living donation (after APOL1 testing is done). The checklist will assess the presence/absence of prescribed counseling practices (fidelity) and a rating of each practice's quality (excellent, very good, good, fair, poor).
  The minimum and maximum values are: 0-12 Higher fidelity scores mean that the post-test counseling discussion exhibited greater fidelity (adherence) to the training program.
  The quality minimum and maximum values are: 1-5 Higher quality scores mean a better quality counseling discussion.

SECONDARY OUTCOMES:
Practical Knowledge and Self-Efficacy in Genetic Counseling | Day 1
  Nephrologists' knowledge and self-efficacy or confidence in their ability to deliver APOL1 counseling will be assessed using a 12-item Likert scale survey. This is the Pre-Test.
  The minimum and maximum values are: 1 to 5 Greater scores reflect greater knowledge or confidence with counseling.
Practical Knowledge and Self-Efficacy in Genetic Counseling | Approximately Day 14
  Nephrologists' knowledge and self-efficacy or confidence in their ability to deliver APOL1 counseling will be assessed using a 12-item Likert scale survey. This is the Post-Test.
  The minimum and maximum values are: 1 to 5 Greater scores reflect greater knowledge or confidence with counseling.
Acceptability of Intervention Measure (AIM) | Approximately Day 21
  This 4-item Likert scale will assess nephrologists' perceptions of the acceptability of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased acceptability of the intervention.
Acceptability of Intervention Measure (AIM) | Approximately Month 2
  This 4-item Likert scale will assess nephrologists' perceptions of the acceptability of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased acceptability of the intervention.
Acceptability of Intervention Measure (AIM) | Approximately Month 12
  This 4-item Likert scale will assess nephrologists' perceptions of the acceptability of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased acceptability of the intervention.
Intervention Appropriateness Measure (IAM) | Approximately Day 21
  This 4-item Likert scale will assess nephrologists' perceptions of the appropriateness of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased perceived appropriateness of the intervention.
Intervention Appropriateness Measure (IAM) | Approximately Month 2
  This 4-item Likert scale will assess nephrologists' perceptions of the appropriateness of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased perceived appropriateness of the intervention.
Intervention Appropriateness Measure (IAM) | Approximately Month 12
  This 4-item Likert scale will assess nephrologists' perceptions of the appropriateness of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased perceived appropriateness of the intervention.
Feasibility of Intervention Measure (FIM) | Approximately Day 21
  This 4-item Likert scale will assess nephrologists' perceptions of the feasibility of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased perceived appropriateness of the intervention.
Feasibility of Intervention Measure (FIM) | Approximately Month 2
  This 4-item Likert scale will assess nephrologists' perceptions of the feasibility of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased perceived appropriateness of the intervention.
Feasibility of Intervention Measure (FIM) | Approximately Month 12
  This 4-item Likert scale will assess nephrologists' perceptions of the feasibility of the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 5 Higher scores indicate increased perceived appropriateness of the intervention.
Clinical Sustainability Assessment Tool (CSAT) | Approximately Month 36
  This 9-item Likert scale will assess nephrologists' perceptions of the sustainability of delivering APOL1 counseling according to the APOL1 counseling training program.
  The minimum and maximum values are: 1 to 7 Higher scores indicate higher capacity for sustainability.

OTHER OUTCOMES:
Racial attributes in clinical evaluation (RACE) scale | Day 1
  This 8-item survey will assess the degree to which nephrologists report using race in their clinical decision making processes.
  The minimum and maximum values are: 0 to 28 Higher scores mean greater use of race in clinical decision-making.
Racial attributes in clinical evaluation (RACE) scale | Approximately Day 14
  This 8-item survey will assess the degree to which nephrologists report using race in their clinical decision making processes.
  The minimum and maximum values are: 0 to 28 Higher scores mean greater use of race in clinical decision-making.
Genetic variation knowledge assessment index (GKAI) | Day 1
  This 8-item survey will assess nephrologists' scientific knowledge of human genetic variation.
  The minimum and maximum values are: 0 to 6 Higher scores mean greater knowledge of genetic variation.
Genetic variation knowledge assessment index (GKAI) | Approximately Day 14
  This 8-item survey will assess nephrologists' scientific knowledge of human genetic variation.
  The minimum and maximum values are: 0 to 6 Higher scores mean greater knowledge of genetic variation.
Health Professionals Beliefs about Race (HPBR) scale | Day 1
  This 9-item survey will assess nephrologists' beliefs about the relationship between race and genetics in terms of race as a biological phenomenon, and the clinical importance of race.
  The scale is scored as two domains: HPBR-Biological domain (contains 4 items that are summed) and HPBR-Clinical domain (contains 3 items that are summed)
  Min-Max: 4 - 20 Biological Domain Min-Max: 3-15 Clinical Domain
  Higher scores indicate greater beliefs about relationships between genetics and race.
Health Professionals Beliefs about Race (HPBR) scale | Approximately Day 14
  This 9-item survey will assess nephrologists' beliefs about the relationship between race and genetics in terms of race as a biological phenomenon, and the clinical importance of race.
  The scale is scored as two domains: HPBR-Biological domain (contains 4 items that are summed) and HPBR-Clinical domain (contains 3 items that are summed)
  Min-Max: 4 - 20 Biological Domain Min-Max: 3-15 Clinical Domain
  Higher scores indicate greater beliefs about relationships between genetics and race.
Barriers and Facilitators to APOL1 testing Implementation | Approximately Day 21
  The Consolidated Framework for Implementation Research Interview guide will be used to assess nephrologists' perceived facilitators and barriers, organizational capacity, and adaptations to the APOL1 testing and counseling program
  This is a qualitative interview guide, thus, there is no minimum or maximum value to be obtained.
Barriers and Facilitators to APOL1 testing Implementation | Approximately Month 3
  The Consolidated Framework for Implementation Research Interview guide will be used to assess nephrologists' perceived facilitators and barriers, organizational capacity, and adaptations to the APOL1 testing and counseling program
  This is a qualitative interview guide, thus, there is no minimum or maximum value to be obtained.
Barriers and Facilitators to APOL1 testing Implementation | Approximately Month 25
  The Consolidated Framework for Implementation Research Interview guide will be used to assess nephrologists' perceived facilitators and barriers, organizational capacity, and adaptations to the APOL1 testing and counseling program
  This is a qualitative interview guide, thus, there is no minimum or maximum value to be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa J Gordon, PhD, MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Medstar Georgetown Transplant Institute, Washington D.C., District of Columbia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith JD, Agrawal A, Wicklund C, Duquette D, Friedewald J, Rasmussen LV, Gacki-Smith J, Tandon SD, Muhammad LN, Yancy CW, Dong S, Cooper M, Gilbert A, Shetty A, Gordon EJ. Implementation of a culturally competent APOL1 genetic testing programme into living donor evaluation: A two-site, non-randomised, pre-post trial design. BMJ Open. 2023 May 15;13(5):e067657. doi: 10.1136/bmjopen-2022-067657. PMID 37188469